CLINICAL TRIAL: NCT04231695
Title: Extracorporeal Cytokine Removal in Patients With Septic Shock in an Adult Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Jose Maria Cullen (Other Government)
Responsible Party: Principal Investigator, Rafael Avila, Rafael Avila ( PI), Hospital Jose Maria Cullen
Other Study IDs: Cytokine
Record Dates: First submitted 2019-12-28; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Septic Shock
Keywords: septic shock; MODS; hemoperfusion; CRRT; ECMO
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Goals Primary: compare changes in norepinephrine requirements before and after hemoperfusion (HP) treatment.

Secondary: demonstrate the decrease in levels of IL-6 , assess the total and individual change of SEQUENTIAL ORGAN FAILURE ASSESSMENT (SOFA), establish the resolution of shock , clearance of lactate , and mortality at discharge from INTENSIVE CARE UNIT (ICU), at 30 and 60 days.

DETAILED DESCRIPTION:
The study will take place at UTI Dr. José María Cullen Hospital in the city of Santa Fe. An observational study will be carried out in adult patients with septic shock (according to the definition of Sepsis-3), presenting hypotension, requiring vasopressors to maintain a mean arterial pressure (MAP) of 65 mmHg, blood lactate> 2 mmol / L, after adequate resuscitation with fluids and in need of extracorporeal membrane oxygenation (Extracorporeal Membrane Oxygenation, ECMO), Renal Replacement Therapy (TRR) ( which may be continuous (Continuous Renal Replacement Therapy (CRRT)) or Extended Slow Daily Dialysis (SLEDD) or both, added to the hemoperfusion (HP) treatment.

The study was designed by the authors, without receiving any input from companies.

Patients will be treated according to The Surviving Sepsis Campaign 2016 recommendations: identification and control of the infectious focus (surgery). It will begin with antibiotics as soon as possible, resuscitation with crystalloids at 30 mL / kg in case of hypotension and continue according to assessment of dynamic and static parameters (EV 1000, Swan Ganz, central venous pressure and echocardiography, used at the discretion of attending physician). Noradrenaline will be administered to maintain a MAP ≧ 65 mmHg. Dobutamine will be indicated if the minute volume <3.0 L / min / m2. According to our practice, adrenaline will be added if the dose of norepinephrine exceeds 2 μg / kg / min. In addition, 100 mg of hydrocortisone will be administered every 8 hours.

In case of requiring TRR for AKI, continuous vein-venous hemodiafiltration will be started using Prismaflex or Amplya equipment with a dose of 35 mL / kg / h, at a 1: 1 ratio, the replacement solution / dialysate solution, with AN ST 1.5 filter, HF 1.4 or HFT 1.4 or 1.7 or 2.2 with citrate as an anticoagulation method. In the case of ECMO, anticoagulation will be performed with heparin, according to the standardized practice of the service.

Treatment with HA 330 cartridges: Hemoperfusion treatment will be initiated as soon as possible, no later than 12 hours after the diagnosis of septic shock. An 8-hour treatment will be indicated for 2 (two) consecutive days. Prior to using the cartridge, 12,500 units of sodium heparin will be placed inside through the hole located in the upper region. During the next 30 minutes, it will be necessary to rotate it so that heparin is distributed throughout its interior. After 30 minutes, a physiological solution should be washed (a total of 2000 mL, with an infusion pump or by gravity pump) in order to remove the heparin, and in turn, avoid the formation of bubbles or air accumulation. After this step it is ready to be used, either for isolated HP therapies or in association with other therapies (SLEDD, ECMO, CRRT )

Data collection: For each patient who enters the protocol, a record will be completed with the data from the sampling, date and time of extraction, with the results of IL-6 and PCT and with the clinical data. The latter will be:

* age
* sex
* preexisting diseases
* infectious focus
* community or acquired sepsis
* positive crops
* SOFA score (daily for 7 (seven) days)
* APACHE II (upon admission and before starting HP treatment)
* IL-6 (as admission criteria and before and after each treatment)
* procalcitonin (PCT) on admission and on days 5-7
* lactate (before and after treatment with HP and daily for 7 (seven) days)
* additional laboratory: blood count, hepatogram, urea, creatinine, coagulogram, norepinephrine / adrenaline / IDI dose
* antibiotic dosing (according to the established sampling scheme)
* administered volume of fluids (daily for 7 (seven) days
* requirement of TRR and ECMO.

Informed consent will be obtained for each patient who enters the protocol for participation Samples will be taken at predetermined times for 48-72 hours following the established procedure.

ELIGIBILITY:
Inclusion Criteria:

1.> 18 years 2. Diagnosis of septic shock (according to sepsis-3 definition) 3. Dose of norepinephrine ≧ 0.4 μg / kg / min 4. Plasma levels of IL-6> 900 pg / mL 5. Procalcitonin (PCT) ≧ 2 ng / mL 6. Need for renal replacement therapies or ECMO

-

Exclusion Criteria:

1. Neoplastic disease with or without treatment
2. Pregnant or lactating women (human chorionic gonadotrophin (hCG) test will be performed on potential patients before recruiting for treatment) -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An observational study will be carried out in adult patients with septic shock (according to the definition of Sepsis-3), presenting hypotension, requiring vasopressors to maintain a mean arterial pressure (MAP) of 65 mmHg, blood lactate> 2 mmol / L, after adequate fluid resuscitation and in need of extracorporeal membrane oxygenation (Extracorporeal Membrane Oxygenation, ECMO), Renal Replacement Therapy (TRR) (which may be continuous (Continuous Renal Replacement Therapy (CRRT)) or Extended Slow Daily Dialysis ( Slow Extended Dialy Dialysis (SLEDD)) or both, added to the hemoperfusion (HP) treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
changes in norepinephrine requirements meassured in micrograms/kg/ min ( gamma) before and after hemoperfusion (HP) treatment. | 8 hours
  we will meassure norepinephrine requirements by placing arterial monitoring during hemoperfusion procedure

SECONDARY OUTCOMES:
levels of IL-6 | 8 hours
  measured by electrochemiluminescence ( picograms/ mililiter)
changes of Sequential Organ Failure Assessment ( SOFA) | 8 hours
  meassured by scale from 0 to 24 where the highest value is worst
concentration of lactate clearence | 8 hours
  (initial lactate - lactate at the end of treatment) / initial lactate x 100
mortality at discharge from UTI | 7 days; 30 days , 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dr Jose Maria Cullen, Santa Fe, Argentina